CLINICAL TRIAL: NCT06539377
Title: Living Donor Liver Transplantation for Neoadjuvant Treated, Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: Living Donor Liver Transplantation for Intrahepatic Cholangiocarcinoma
Acronym: LIVINCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Responsible Party: Principal Investigator, Falk Rauchfuß, Prof. Dr. med. Falk Rauchfuß, Sectio head liver transplantation, Principal investigator, Jena University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-3430-BO
Record Dates: First submitted 2024-07-30; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Living Donor Liver Transplantation; Liver Transplantation; Neoadjuvant Therapy
Keywords: intrahepatic cholangiocarcinoma; living donor liver transplantation; neoadjuvant therapy; SIRT
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Intervention Model Description: Curative treatment of unresectable intrahepatic cholangiocarcinoma via living donor donation and one- or two-staged hepatectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Living donor liver transplantation (Experimental): The evaluation tests prior the transplantation will be performed following the standard protocol for the evaluation of a waiting list applicants prior liver transplantation. The aim of this procedure is to rule out any significant co-morbidities (e.g. cardiologic diseases, other malignancies) which would preclude liver transplantation.
  After successful evaluation of the recipient and waiting list registration with Eurotransplant, the AB0-compatible donor will be evaluated as well according to a center-specific protocol.
  For a local control of the tumor, an additional local-ablative therapy (SIRT) is mandatory.
  Interventions: Procedure: Living donor liver transplantation

INTERVENTIONS:
Procedure: Living donor liver transplantation — Liver transplantation from living donor donation (SII/III as left-lateral donation during a "two stage"-procedure or left lobe donation or right lobe donation) in patients with unresectable intrahepatic cholangiocarcinoma.

SUMMARY:
This study is supposed to make liver transplantation available for treatment in well selected patients suffering from non-resectable intrahepatic cholangiocarcinoma. Donor organ shortage is currently the main problem for organ transplantation world-wide. Thus, the particular indication "non-resectable intrahepatic cholangiocarcinoma" is currently excluded in terms of transplantation. Given those circumstances, transplantation via living donation might be the best option. This procedure does not reduce the deceased donor organ supply because living donation is the primary treatment option in these patients (not subsidiary).

DETAILED DESCRIPTION:
Intrahepatic cholangiocarcinoma (iCCA) is classified among primary liver tumors and has demonstrated a consistently increasing incidence in recent years. Due to the poor long-term survival rates reported in older studies, liver transplantation continues to be a contraindication in the curative treatment of iCCA. The persistent shortage of organs also necessitates that each new indication for transplantation be carefully evaluated and critically scrutinized. Currently, partial resection remains the preferred treatment modality, although at diagnosis, only approximately 20% of cases are amenable to this approach. Post-partial resection, the five-year survival rate is observed to be between 20-34%. In cases of irresectability, palliative chemotherapy often remains the only option, typically associated with a poor prognosis. Numerous studies have demonstrated that long-term outcomes following liver transplantation for iCCA have evolved and improved over the years. In a meta-analysis by Ziogas et al., data from a total of 18 studies (involving 355 patients) and one registry study (385 patients) were analyzed. The pooled 1-, 3-, and 5-year survival rates were 75%, 56%, and 42%, respectively. Meanwhile, the pooled 1-, 3-, and 5-year recurrence-free survival rates were 70%, 49%, and 38%, with an overall recurrence rate of 43%. A potential reason for this marked improvement may be attributed to the introduction of neoadjuvant therapy. Studies by Hu et al. and Lunsford et al. have demonstrated that the utilization of neoadjuvant therapy is associated with significantly improved survival outcomes. The study aims to conduct a prospective, non-randomized study (LIVINCA) to further explore the effects of living-donor liver transplantation in the treatment of unresectable neoadjuvant treated (chemotherapy AND selective internal radiotherapy) intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* non-resectable intrahepatic cholangiocarcinoma (either for localization / distribution of the carcinoma or for estimated function of the liver in case of liver fibrosis / cirrhosis)
* biopsy proven grading G1 / G2
* in case of mixed hepatocellular carcinoma / cholangiocarcinoma, the cholangiocarcinoma also must have a grading of G1 / G2
* response to chemotherapy in terms of stable or regressive disease (imaging studies, tumor marker CA19-9, any chemotherapy regime allowed, a local-ablative therapy in means of a SIRT is mandatory
* peritoneal carcinosis / extrahepatic spread ruled out in PET-CT and/or MRT/CT and, at latest, during exploration
* age ≥ 18
* blood-group compatible living donor available
* in female patients: negative pregnancy test
* written informed consent before study enrolment of donor and recipient (all other procedures are clinical routine procedures in the management of these patients)

Exclusion Criteria:

* extrahepatic tumor/metastases
* G3 tumors
* progress under neoadjuvant treatment according to the RECIST-criteria
* pregnancy or breastfeeding
* patients unwilling to consent to saving and propagation of pseudonymized medical data for study reasons
* general contraindications for liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2030-10-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
Five year overall survival | Five years
  Survival from time of transplantation to time of death or last follow up

SECONDARY OUTCOMES:
Recurrence-free survival | Five years
  Survival from time of transplantation to time of death or first evidence of recurrence to disease
Donor and Recipient morbidity | Five years
  Donor and Recipient morbidity (both according to the Clavien-Dindo classification)

CONTACTS AND LOCATIONS:
Overall Officials: Utz Settmacher, Prof, Study Director — Jena University Hospital; Falk Rauchfuss, Prof, Study Director — Jena University Hospital; Laura Schwenk, MD, Study Director — Jena University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldaracena N, Gorgen A, Sapisochin G. Current status of liver transplantation for cholangiocarcinoma. Liver Transpl. 2018 Feb;24(2):294-303. doi: 10.1002/lt.24955. PMID 29024405
- [Background] Ziogas IA, Giannis D, Economopoulos KP, Hayat MH, Montenovo MI, Matsuoka LK, Alexopoulos SP. Liver Transplantation for Intrahepatic Cholangiocarcinoma: A Meta-analysis and Meta-regression of Survival Rates. Transplantation. 2021 Oct 1;105(10):2263-2271. doi: 10.1097/TP.0000000000003539. PMID 33196623
- [Background] Chan KM, Tsai CY, Yeh CN, Yeh TS, Lee WC, Jan YY, Chen MF. Characterization of intrahepatic cholangiocarcinoma after curative resection: outcome, prognostic factor, and recurrence. BMC Gastroenterol. 2018 Dec 4;18(1):180. doi: 10.1186/s12876-018-0912-x. PMID 30514231
- [Background] Lunsford KE, Javle M, Heyne K, Shroff RT, Abdel-Wahab R, Gupta N, Mobley CM, Saharia A, Victor DW, Nguyen DT, Graviss EA, Kaseb AO, McFadden RS, Aloia TA, Conrad C, Li XC, Monsour HP, Gaber AO, Vauthey JN, Ghobrial RM; Methodist-MD Anderson Joint Cholangiocarcinoma Collaborative Committee (MMAJCCC). Liver transplantation for locally advanced intrahepatic cholangiocarcinoma treated with neoadjuvant therapy: a prospective case-series. Lancet Gastroenterol Hepatol. 2018 May;3(5):337-348. doi: 10.1016/S2468-1253(18)30045-1. Epub 2018 Mar 13. PMID 29548617
- [Background] McMillan RR, Javle M, Kodali S, Saharia A, Mobley C, Heyne K, Hobeika MJ, Lunsford KE, Victor DW 3rd, Shetty A, McFadden RS, Abdelrahim M, Kaseb A, Divatia M, Yu N, Nolte Fong J, Moore LW, Nguyen DT, Graviss EA, Gaber AO, Vauthey JN, Ghobrial RM. Survival following liver transplantation for locally advanced, unresectable intrahepatic cholangiocarcinoma. Am J Transplant. 2022 Mar;22(3):823-832. doi: 10.1111/ajt.16906. Epub 2021 Dec 27. PMID 34856069